CLINICAL TRIAL: NCT00311597
Title: A Phase I/II Dose-Escalation/Efficacy Study of Palliative Extracranial Radiosurgery Using the Elektra Stereotactic Body Frame System
Brief Title: Extracranial Stereotactic Radiosurgery in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000466064; CCCWFU-99502; CCCWFU-BG02-187
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single fractionated radiation adjusted for tumor size (Experimental): Single fractionated radiation adjusted for volume of tumor tissue encompassed by desired isodose line
  Interventions: Procedure: Radiosurgery

INTERVENTIONS:
Procedure: Radiosurgery — single fractionated radiation therapy

SUMMARY:
RATIONALE: Extracranial stereotactic radiosurgery may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This phase I/II trial is studying the side effects and best dose of extracranial stereotactic radiosurgery and to see how well it works in treating patients with solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Establish the maximum tolerated dose (MTD) of extracranial stereotactic radiosurgery in patients with isolated tumors. (Phase I)
* Determine the minimum dose required for local control. (Phase II)

Secondary

* Determine the radiographic response rate.
* Determine the median time to progression of the treated tumor.
* Evaluate the toxicity of treatment.
* Evaluate the cause of death.

OUTLINE: This is a phase I dose-escalation study followed by a phase II open-label study. Patients are stratified according to tumor size.

* Phase I: Patients undergo stereotactic radiosurgery to one lesion. Cohorts of 3-6 patients undergo escalating doses of stereotactic radiosurgery until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 33% of patients experience dose-limiting toxicity within 3 months of treatment.
* Phase II: Patients undergo stereotactic radiosurgery to one lesion at the MTD or at the dose at which local control at 3 months is ≥ 80%, as determined in phase I.

After completion of study treatment, patients are followed at 1 month, 3 months, and then every 3 months thereafter.

PROJECTED ACCRUAL: At least 48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Presence of well-circumscribed tumor on contrast-enhanced CT scan or MRI

  * Maximum diameter of 6 cm

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 3 months
* Not pregnant
* Fertile patients must use effective contraception
* Negative pregnancy test
* Must be able to tolerate CT scan or MRI contrast

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since prior chemotherapy or immunotherapy
* No prior treatment on this study
* No chemotherapy or immunotherapy during and for 4 weeks after completion of study treatment
* No concurrent external-beam radiotherapy overlapping with the radiosurgically-treated volume (including low-dose regions)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2002-06 (Actual); Primary Completion 2007-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose for up to 90 days after completion of study treatment | day 1 through 90
Minimum dose required for local control as assessed by RECIST one-dimensional criterion and volumetric analysis for 90 days after completion of study treatment | day 1 through 90

SECONDARY OUTCOMES:
Median time to progression of treated tumor for up to 2 years | day 1 to 2 years
Toxicity as assessed by NCI Common Toxicity Criteria (CTC) version 2.0 for up to 90 days after completion of study treatment | day 1 through 90
Cause of death as assessed by medical records and autopsy at time of death | variable, survival of the patient

CONTACTS AND LOCATIONS:
Overall Officials: James Urbanic, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Stieber VW, Hinson W, Kearns W, et al.: A phase I/II dose-escalation/efficacy study of palliative stereotactic body radiosurgery, including bioanatomic imaging to assess response. [Abstract] Int J Radiat Oncol Biol Phys 60 (1 Suppl 1): A-2381, S563-4, 2004.